CLINICAL TRIAL: NCT01865526
Title: Effects of the 6-point Diet on the Metabolic Control, the Compliance and the Nutritional Status of CKD Patients Stage 3b-5
Brief Title: Efficacy of the 6-point Diet
Acronym: PIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Eleonora Riccio, MD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PIS; Carlo Romano (Other: Ethic commettee)
Record Dates: First submitted 2013-05-24; First posted 2013-05-31 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2012-12

CONDITIONS: Chronic Kidney Disease
Keywords: Chronic kidney disease; Low protein diet; CKD stage 3b-5
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Diet, Protein-Restricted

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Low protein diet (Active Comparator): The patients of this group received a classical low protein diet (LPD),according to their desired body weight (DBW), obtained by multiplying the squared value of the height times a reference body mass index (BMI) value of 23. LPD were individually prepared and explained to the patients by a dedicated dietician and contained at least 30 kcal/kg/day (25 in overweight patients), with a dietary sodium intake restricted to 2.5 g/day.
  Interventions: Dietary Supplement: Low protein diet
- Six point diet (Experimental): These patients were assigned to receive the 6-points-diet, and were given by the Nephrologist the list of six items indicating how to modify their dietary habits; all the items were thoroughly explained and discussed with the patients
  Interventions: Dietary Supplement: Six point diet

INTERVENTIONS:
Dietary Supplement: Six point diet — The 6-point diet is a list of six items indicating how to modify their dietary habits:
  1. Do not add salt at table and for cooking;
  2. Food to avoid: any kind of salami, sausages, cheese and dairy products or canned food;
  3. Replace noodle or bread with special no-protein food;
  4. The second course (meat, fish and eggs) are allowed once a day in the usual quantity;
  5. 4-5 servings/day of fruits or vegetables are suggested;
  6. Once or twice a week the main course may be of "normal" noodle with legumes instead of the second course, with fruit and vegetables.
  Arms: Six point diet
Dietary Supplement: Low protein diet — Classical low-protein diet prescribed according to the patients' desired body weight (DBW), obtained by multiplying the squared value of the height times a reference BMI value of 23. These diets contained at least 30 kcal/kg/day (25 in overweight patients), with a dietary sodium intake restricted to 2.5 g/day.
  Arms: Low protein diet

SUMMARY:
The dietary restriction of proteins and sodium is a cornerstone in the treatment of chronic kidney disease (CKD) and of its metabolic consequences. Dietary adjustments in CKD are complex and the patients' compliance is very low. A dietary interview method is a validated instrument to evaluate the patients' compliance; however, it the presence of a dedicated dietitians. For these reasons, and because of the absence of dedicated dietitians in many nephrology centres, it is usual practice to give standard low protein diets to CKD patients not on dialysis.

Aim of this study was to verify if few simple tips were able to reduce protein, phosphate and sodium intake in patients with CKD, as compared to the practice of giving a low protein diet elaborated by a renal dietitian.

DETAILED DESCRIPTION:
The dietary restriction of proteins and sodium is a cornerstone in the treatment of chronic kidney disease (CKD) and of its metabolic consequences. In fact, a reduced protein intake decreases load on remaining nephrons, reduces signs and symptoms of uraemia, lessens the accumulation of waste metabolic products and oxidant stress, improves insulin-resistance and lipid profile, ameliorates proteinuria, additives effects of angiotensin-converting-enzyme inhibitors, and decreases likelihood of patients death or delays initiation of dialysis by 40%.

Dietary adjustments in subjects with chronic renal failure are complex because multiple nutrient modifications are required and changes in lifestyle must be maintained for years. Furthermore, low-protein diet is considered tedious, unpalatable and difficult to achieve. This has an obvious negative influence on the quality of life of patients and makes their adherence to the new therapeutic prescriptions more difficult. In fact, the difficulty to reach patients' compliance is well known. There is ample evidence that poor adherence is considered a critical barrier to treatment success and remains one of the leading challenges to healthcare professionals. Few data are available in clinical practice concerning the patients' compliance to low protein diet. A dietary interview method is a validated instrument to evaluate the practice and routines related to the assessment of nutrient intake in nondialyzed CKD patients and to obtain the patients' compliance. However, the interview requires the presence of a dedicated dietitian and a lot of his time.

For these reasons, and because of the absence of dedicated dietitians in many nephrology centres, it is usual practice to give standard low protein diets to CKD patients not on dialysis.

Aim of this study was to verify if few simple tips were able to reduce protein, phosphate and sodium intake in patients with CKD, as compared to the practice of giving a low protein diet elaborated by a renal dietitian.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years
* a basal value of estimated GFR (eGFR) < 45 ml/min/1,73 m2, that had to remain stable during 3 consecutive controls (eGFR variability <15% along 1 month)

Exclusion Criteria:

* unstable renal function,
* inability to perform correct 24-hours urine collections,
* presence of malignancies,
* treatment with immunosuppressive drugs,
* pregnancy,
* congestive heart failure (NYHA class III-IV),
* proteinuria >3,5 g/24 hours

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2010-03; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Effect on renal disease progression | 6 months
  Evaluation of modification of GFR and proteinuria
Effect on metabolic control | 6 months
  Evaluation of the modifications of serum urea nitrogen, sodium, potassium, phosphate, bicarbonate, parathormone , urinary urea nitrogen, phosphate, potassium, sodium, protein and phosphate intake
Effect on nutritional status | 6 months
  Evaluation of modifications of total protein, albumin, C-reactive protein, body weight, BMI
Effect on patients'compliance to the dietetic therapy | 6 months
  The compliance was defined by a constant protein intake between 0.7 and 0.9 g/kg B.W. throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: eleonora riccio, md, Principal Investigator — Federico II University
Locations (1):
- federico II university, department of nephrology, Naples, Naples, Italy

REFERENCES:
- [Derived] Pisani A, Riccio E, Bellizzi V, Caputo DL, Mozzillo G, Amato M, Andreucci M, Cianciaruso B, Sabbatini M. 6-tips diet: a simplified dietary approach in patients with chronic renal disease. A clinical randomized trial. Clin Exp Nephrol. 2016 Jun;20(3):433-42. doi: 10.1007/s10157-015-1172-5. Epub 2015 Oct 9. PMID 26453483